CLINICAL TRIAL: NCT01641237
Title: The Effect of Fluoride in an Experimental Dentifrice on Remineralization of Erosive Lesions In-Situ
Brief Title: Effect of Fluoride in a Dentifrice on Remineralization of Erosive Lesions
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: RH01299
Record Dates: First submitted 2012-07-12; First posted 2012-07-16 (Estimated); Results first posted 2013-07-31 (Estimated); Last update posted 2014-07-24 (Estimated); Status verified 2014-06

CONDITIONS: Enamel Erosion
MeSH Terms: interventions — Sodium Fluoride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Low ppm fluoride dentifrice (Experimental): Low ppm fluoride as sodium fluoride in a silica base dentifrice
  Interventions: Drug: sodium fluoride
- Medium ppm fluoride dentifrice (Experimental): Medium ppm fluoride as sodium fluoride in a silica base dentifrice
  Interventions: Drug: sodium fluoride
- High ppm fluoride dentifrice (Experimental): High ppm fluoride as sodium fluoride in a silica base dentifrice
  Interventions: Drug: sodium fluoride
- No fluoride dentifrice (Placebo Comparator): no added fluoride in a silica base dentifrice
  Interventions: Drug: no added fluoride in a silica base

INTERVENTIONS:
Drug: sodium fluoride — fluoride as sodium fluoride
  Arms: High ppm fluoride dentifrice; Low ppm fluoride dentifrice; Medium ppm fluoride dentifrice
Drug: no added fluoride in a silica base — no added fluoride
  Arms: No fluoride dentifrice

SUMMARY:
The proposed study will evaluate the performance of fluoride delivered from a new dentifrice formulation without potassium nitrate. It will also evaluate the dose-response to fluoride by testing four dentifrices covering a range of sodium fluoride concentration.

ELIGIBILITY:
Inclusion Criteria:

* intact maxillary dental arch suitable to retain a palatal appliance, an intact mandibular dental arch and a stimulated/unstimulated saliva flow rate of ≥ 0.8 milliliter/minute (ml/min) and ≥ 0.2 ml/min respectively.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2012-03; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- Indiana University School of Dentistry, Indianapolis, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at the clinical site.
Pre-assignment Details: A total of 72 participants were screened, and 62 were randomized into the study. 9 participants did not meet the study criteria and 1 withdrew consent. A washout non-fluoridated toothpaste was used for 2 days prior treatment. In-situ appliances were prepared for participants to fit enamel specimens.
Groups:
- Sodium Fluoride (NaF) Dentifrice,1426 Parts Per Million(Ppm)F: Participants were fitted with enamel specimen appliance in the palatal surface 5 minutes before treatment initiation. Participants brushed their teeth for one timed minute with 1.5 grams (g) ± 0.1g of NaF toothpaste (1426 ppmF) and expectorated. The direct contact between palatal appliance and toothbrush was avoided.
- NaF Dentifrice (1150ppmF): Participants were fitted with enamel specimen appliance in the palatal surface 5 minutes before treatment initiation. Participants brushed their teeth for one timed minute with 1.5 g ± 0.1g of NaF toothpaste (1150 ppmF) and expectorated. The direct contact between palatal appliance and toothbrush was avoided.
- NaF Dentifrice (250ppmF): Participants were fitted with enamel specimen appliance in the palatal surface 5 minutes before treatment initiation. Participants brushed their teeth for one timed minute with 1.5 g ± 0.1g of NaF toothpaste (250 ppmF) and expectorated. The direct contact between palatal appliance and toothbrush was avoided.
- Placebo Dentifrice (0ppmF): Participants were fitted with enamel specimen appliance in the palatal surface 5 minutes before treatment initiation. Participants brushed their teeth for one timed minute with 1.5 g ± 0.1g of placebo toothpaste (0 ppmF) and expectorated. The direct contact between palatal appliance and toothbrush was avoided.
Period: Period I
Arm/Group | Sodium Fluoride (NaF) Dentifrice,1426 Parts Per Million(Ppm)F | NaF Dentifrice (1150ppmF) | NaF Dentifrice (250ppmF) | Placebo Dentifrice (0ppmF)
Started | 16 | 16 | 15 | 15
Completed | 16 | 16 | 15 | 15
Not Completed | 0 | 0 | 0 | 0
Period: Period II
Arm/Group | Sodium Fluoride (NaF) Dentifrice,1426 Parts Per Million(Ppm)F | NaF Dentifrice (1150ppmF) | NaF Dentifrice (250ppmF) | Placebo Dentifrice (0ppmF)
Started | 15 (Due to crossover design, different set of participants entered Period 2) | 16 (Due to crossover design, different set of participants entered Period 2) | 16 (Due to crossover design, different set of participants entered Period 2) | 15 (Due to crossover design, different set of participants entered Period 2)
Completed | 14 | 16 | 16 | 15
Not Completed | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0
Period: Period III
Arm/Group | Sodium Fluoride (NaF) Dentifrice,1426 Parts Per Million(Ppm)F | NaF Dentifrice (1150ppmF) | NaF Dentifrice (250ppmF) | Placebo Dentifrice (0ppmF)
Started | 16 (Due to crossover design, different set of participants entered Period 3) | 14 (Due to crossover design, different set of participants entered Period 3) | 15 (Due to crossover design, different set of participants entered Period 3) | 16 (Due to crossover design, different set of participants entered Period 3)
Completed | 15 | 14 | 15 | 16
Not Completed | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0
Period: Period IV
Arm/Group | Sodium Fluoride (NaF) Dentifrice,1426 Parts Per Million(Ppm)F | NaF Dentifrice (1150ppmF) | NaF Dentifrice (250ppmF) | Placebo Dentifrice (0ppmF)
Started | 15 (Due to crossover design, different set of participants entered Period 4) | 15 (Due to crossover design, different set of participants entered Period 4) | 15 (Due to crossover design, different set of participants entered Period 4) | 15 (Due to crossover design, different set of participants entered Period 4)
Completed | 15 | 15 | 15 | 15
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Randomized Participants: All randomized participants who received at least one dose of the study treatments.
Arm/Group | All Randomized Participants
Number analyzed (Participants) | 62
Age, Continuous [Mean (Standard Deviation); unit: Years] | 36.7 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35
  Male | 27

OUTCOME MEASURES:

1. Primary Outcome: Percentage Surface Microhardness Recovery (%SMHR) Dose Response Relationship
Description: SMHR test was used to assess the changes in mineralization status of enamel specimens using a Wilson 2100 Hardness tester. SMHR was determined by measuring the length of the indentations of enamel specimens. An increase in the indentation length compared to the baseline indicates softening while decrease in the indentation length represents rehardening of enamel surface. Percent SMHR was calculated from indentation values of enamel specimens at baseline (B), after in-situ hardening (R) and after first erosive challenge (E1) using formula: [(E1-R)/ (E1-B)]*100.
Time Frame: Baseline to 4 hours
Population: Per protocol population: All randomized participants who received at least one study product, had one efficacy assessment and did not have any protocol violations deemed to affect efficacy. Missing values were not imputed.
Measure: Mean (Standard Error); unit: %SMHR
Groups:
- NaF Dentifrice (1426 ppmF): Participants were fitted with enamel specimen appliance in the palatal surface 5 minutes before treatment initiation. Participants brushed their teeth for one timed minute with 1.5 g ± 0.1g of NaF toothpaste (1426 ppmF) and expectorated. The direct contact between palatal appliance and toothbrush was avoided.
- NaF Dentifrice (1150 ppmF): Participants were fitted with enamel specimen appliance in the palatal surface 5 minutes before treatment initiation. Participants brushed their teeth for one timed minute with 1.5 g ± 0.1g of NaF toothpaste (1150 ppmF) and expectorated. The direct contact between palatal appliance and toothbrush was avoided.
- NaF Dentifrice (250 ppmF): Participants were fitted with enamel specimen appliance in the palatal surface 5 minutes before treatment initiation. Participants brushed their teeth for one timed minute with 1.5 g ± 0.1g of NaF toothpaste (250 ppmF) and expectorated. The direct contact between palatal appliance and toothbrush was avoided.
- Placebo Dentifrice (0 ppmF): Participants were fitted with enamel specimen appliance in the palatal surface 5 minutes before treatment initiation. Participants brushed their teeth for one timed minute with 1.5 g ± 0.1g of placebo toothpaste (0 ppmF) and expectorated. The direct contact between palatal appliance and toothbrush was avoided.
Arm/Group | NaF Dentifrice (1426 ppmF) | NaF Dentifrice (1150 ppmF) | NaF Dentifrice (250 ppmF) | Placebo Dentifrice (0 ppmF)
Number analyzed (Participants) | 61 | 61 | 61 | 60
%SMHR | 30.89 (1.38) | 28.71 (1.38) | 25.28 (1.38) | 21.03 (1.39)
Statistical Analysis 1: Comparison: NaF Dentifrice (1426 ppmF) vs NaF Dentifrice (1150 ppmF) vs NaF Dentifrice (250 ppmF) vs Placebo Dentifrice (0 ppmF); Test for linear dose-response relationship was performed for %SMHR as a function of fluoride concentration; Test type: Superiority or Other; p < 0.0001, ANOVA; Adjusted Mean and SE were calculated from ANOVA model with treatment and period as factors, and subject as a random factor
Statistical Analysis 2: Comparison: NaF Dentifrice (1426 ppmF) vs NaF Dentifrice (1150 ppmF) vs NaF Dentifrice (250 ppmF) vs Placebo Dentifrice (0 ppmF); Test for quadratic dose-response relationship was performed for %SMHR as a function of fluoride concentration; Test type: Superiority or Other; p = 0.3748, ANOVA; [statistical method as in outcome 1, analysis 1]

2. Secondary Outcome: %SMHR
Description: as for outcome 1
Time Frame: Baseline to 4 hours
Population: PP population: All randomized participants who received at least one study product, had one efficacy assessment and did not have any protocol violations deemed to affect efficacy. Missing values were not imputed.
Measure: Mean (Standard Error); unit: %SMHR
Arm/Group | NaF Dentifrice (1426 ppmF) | NaF Dentifrice (1150 ppmF) | NaF Dentifrice (250 ppmF) | Placebo Dentifrice (0 ppmF)
Number analyzed (Participants) | 61 | 61 | 61 | 60
%SMHR | 30.9 (1.38) | 28.7 (1.38) | 25.3 (1.38) | 21.0 (1.39)
Statistical Analysis 1: Comparison: NaF Dentifrice (1426 ppmF) vs NaF Dentifrice (1150 ppmF); Null hypothesis considered treatments in comparison to be equal; Test type: Superiority or Other; p = 0.1898, ANOVA — No adjustment was required for multiple comparisons as the primary comparison was pre-specified; ANOVA with fixed factors for study period and treatment and the subject as random effect; Adjusted Mean Difference = 2.17, 95% CI 2-sided [-1.09 to 5.43] — Difference is first named treatment minus second named treatment such that a positive difference favors the first named treatment
Statistical Analysis 2: Comparison: NaF Dentifrice (1426 ppmF) vs NaF Dentifrice (250 ppmF); Null hypothesis considered no dose-response relationship between %SMHR and fluoride concentration in the dentifrice; Test type: Superiority or Other; p = 0.0009, ANOVA — No adjustment was required for multiple comparisons as the primary comparison was pre-specified; ANOVA with fixed factors for study period and treatment and the subject as random effect; Adjusted Mean Difference = 5.60, 95% CI 2-sided [2.35 to 8.86] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: NaF Dentifrice (1150 ppmF) vs NaF Dentifrice (250 ppmF); Null hypothesis considered treatments in comparison to be equal; Test type: Superiority or Other; p = 0.0389, ANOVA — No adjustment was required for multiple comparisons as the primary comparison was pre-specified; ANOVA with fixed factors for study period and treatment and the subject as random effect; Adjusted Mean Difference = 3.43, 95% CI 2-sided [0.18 to 6.68] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 4: Comparison: NaF Dentifrice (1426 ppmF) vs Placebo Dentifrice (0 ppmF); Null hypothesis considered treatments in comparison to be equal; Test type: Superiority or Other; p < 0.0001, ANOVA — No adjustment was required for multiple comparisons as primary comparison was pre-specified; ANOVA with fixed factors for study period and treatment, and subject as random effect; Adjusted Mean Difference = 9.86, 95% CI 2-sided [6.58 to 13.13] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 5: Comparison: NaF Dentifrice (1150 ppmF) vs Placebo Dentifrice (0 ppmF); Null hypothesis considered treatments in comparison to be equal; Test type: Superiority or Other; p < 0.0001, ANOVA — No adjustment was required for multiple comparisons as primary comparison was pre-specified; ANOVA with fixed factors for study period and treatment, and subject as random effect; Adjusted Mean Difference = 7.68, 95% CI 2-sided [4.41 to 10.96] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 6: Comparison: NaF Dentifrice (250 ppmF) vs Placebo Dentifrice (0 ppmF); Null hypothesis considered treatments in comparison to be equal; Test type: Superiority or Other; p = 0.0112, ANOVA — No adjustment was required for multiple comparisons as primary comparison was pre-specified; ANOVA with fixed factors for study period and treatment, and subject as random effect; Adjusted Mean Difference = 4.25, 95% CI 2-sided [0.98 to 7.53] — [estimate comment as in outcome 2, analysis 1]

3. Secondary Outcome: Percentage Relative Erosion Resistance
Description: Changes in mineral content of enamel specimens exposed to dietary erosive challenge were determined by measuring the length of the indentations. Decrease in the indentation length compared to the baseline indicates hardening of enamel surface. Enamel specimens were exposed to second erosion challenge to determine relative erosion resistance which compared the indentations values of enamel specimens at baseline (B), first erosive (E1) and second erosive challenge (E2). Percent relative erosion resistance was calculated by formula: [(E1-E2)/ (E1-B)]*100.
Time Frame: Baseline to 4 hours
Population: as for outcome 2
Measure: Mean (Standard Error); unit: % Relative Erosion Resistance
Arm/Group | NaF Dentifrice (1426 ppmF) | NaF Dentifrice (1150 ppmF) | NaF Dentifrice (250 ppmF) | Placebo Dentifrice (0 ppmF)
Number analyzed (Participants) | 61 | 61 | 61 | 60
% Relative Erosion Resistance | -38.83 (2.75) | -39.75 (2.75) | -50.40 (2.75) | -71.21 (2.77)
Statistical Analysis 1: Comparison: NaF Dentifrice (1426 ppmF) vs NaF Dentifrice (1150 ppmF) vs NaF Dentifrice (250 ppmF) vs Placebo Dentifrice (0 ppmF); Test for linear dose-response relationship was performed for %RER as a function of fluoride concentration; Test type: Superiority or Other; p < 0.0001, ANOVA; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: NaF Dentifrice (1426 ppmF) vs NaF Dentifrice (1150 ppmF) vs NaF Dentifrice (250 ppmF) vs Placebo Dentifrice (0 ppmF); Test for quadratic dose-response relationship was performed for %RER as a function of fluoride concentration; Test type: Superiority or Other; p = 0.0002, ANOVA
Statistical Analysis 3: Comparison: NaF Dentifrice (1426 ppmF) vs Placebo Dentifrice (0 ppmF); Null hypothesis considered no difference between treatments, being compared; Test type: Superiority or Other; p < 0.0001, ANOVA — No adjustment was required for multiple comparisons as primary comparison was pre-specified; ANOVA with fixed factors for study period and treatment, while subject was random effect; Adjusted Mean Difference = 32.38, 95% CI 2-sided [25.18 to 39.59] — Difference was first named treatment minus second named treatment such that a positive difference favors the first named treatment
Statistical Analysis 4: Comparison: NaF Dentifrice (1150 ppmF) vs Placebo Dentifrice (0 ppmF); Null hypothesis considered no difference between treatments, being compared; Test type: Superiority or Other; p < 0.0001, ANOVA — No adjustment was required for multiple comparisons as primary comparison was pre-specified; ANOVA with fixed factors for study period and treatment, while subject was random effect; Adjusted Mean Difference = 31.46, 95% CI 2-sided [24.25 to 38.67] — [estimate comment as in outcome 3, analysis 3]
Statistical Analysis 5: Comparison: NaF Dentifrice (250 ppmF) vs Placebo Dentifrice (0 ppmF); Null hypothesis considered no difference between treatments, being compared; Test type: Superiority or Other; p < 0.0001, ANOVA — No adjustment was required for multiple comparisons as primary comparison was pre-specified; ANOVA with fixed factors for study period and treatment, while subject was random effect; Adjusted Mean Difference = 20.81, 95% CI 2-sided [13.60 to 28.02] — [estimate comment as in outcome 3, analysis 3]
Statistical Analysis 6: Comparison: NaF Dentifrice (1426 ppmF) vs NaF Dentifrice (1150 ppmF); Null hypothesis considered no difference between treatments, being compared; Test type: Superiority or Other; p = 0.8000, ANOVA — No adjustment was required for multiple comparisons as primary comparison was pre-specified; ANOVA with fixed factors for study period and treatment, while subject was random effect; Adjusted Mean Difference = 0.92, 95% CI 2-sided [-6.25 to 8.10] — [estimate comment as in outcome 3, analysis 3]
Statistical Analysis 7: Comparison: NaF Dentifrice (1426 ppmF) vs NaF Dentifrice (250 ppmF); Null hypothesis considered no difference between treatments, being compared; Test type: Superiority or Other; p = 0.0017, ANOVA — No adjustment was required for multiple comparisons as primary comparison was pre-specified; ANOVA with fixed factors for study period and treatment, while subject was random effect; Adjusted Mean Difference = 11.57, 95% CI 2-sided [4.40 to 18.74] — [estimate comment as in outcome 3, analysis 3]
Statistical Analysis 8: Comparison: NaF Dentifrice (1150 ppmF) vs NaF Dentifrice (250 ppmF); Null hypothesis considered no difference between treatments, being compared; Test type: Superiority or Other; p = 0.0038, ANOVA — No adjustment was required for multiple comparisons as primary comparison was pre-specified; ANOVA with fixed factors for study period and treatment, while subject was random effect; Adjusted Mean Difference = 10.65, 95% CI 2-sided [3.48 to 17.81] — [estimate comment as in outcome 3, analysis 3]

4. Secondary Outcome: Enamel Fluoride Uptake (Corrected Data)
Description: Enamel fluoride uptake was determined using the microdrill enamel biopsy technique. The amount of fluoride uptake by enamel was calculated based on amount of fluoride divided by area of the enamel cores. Data analysis was based on corrected data.
Time Frame: Baseline to 4 hours
Population: PP population: All randomized participants who received at least one study product, had one efficacy assessment and did not have any protocol violations deemed to affect efficacy. Missing values were not imputed. Data analysis for this outcome measure was performed based on a correction factor.
Measure: Mean (Standard Error); unit: micrograms*F/centimeters^2
Arm/Group | NaF Dentifrice (1426 ppmF) | NaF Dentifrice (1150 ppmF) | NaF Dentifrice (250 ppmF) | Placebo Dentifrice (0 ppmF)
Number analyzed (Participants) | 61 | 61 | 61 | 60
micrograms*F/centimeters^2 | 3.13 (0.09) | 3.07 (0.09) | 2.09 (0.09) | 1.47 (0.09)
Statistical Analysis 1: Comparison: NaF Dentifrice (1426 ppmF) vs NaF Dentifrice (1150 ppmF) vs NaF Dentifrice (250 ppmF) vs Placebo Dentifrice (0 ppmF); Test for linear dose-response relationship was performed for EFU as a function of fluoride concentration; Test type: Superiority or Other; p < 0.0001, ANOVA; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: NaF Dentifrice (1426 ppmF) vs NaF Dentifrice (1150 ppmF) vs NaF Dentifrice (250 ppmF) vs Placebo Dentifrice (0 ppmF); Test for quadratic dose-response relationship was performed for EFU as a function of fluoride concentration; Test type: Superiority or Other; p = 0.0008, ANOVA; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: NaF Dentifrice (1426 ppmF) vs Placebo Dentifrice (0 ppmF); Null hypothesis considered no difference between treatments, being compared; Test type: Superiority or Other; p < 0.0001, ANOVA — No adjustment was required for multiple comparisons as primary comparison was pre-specified; ANOVA with fixed factors for study period and treatment, while subject was random effect; Adjusted Mean Difference = 1.66, 95% CI 2-sided [1.42 to 1.90] — [estimate comment as in outcome 3, analysis 3]
Statistical Analysis 4: Comparison: NaF Dentifrice (1150 ppmF) vs Placebo Dentifrice (0 ppmF); Null hypothesis considered no difference between treatments, being compared; Test type: Superiority or Other; p < 0.0001, ANOVA — No adjustment was required for multiple comparisons as primary comparison was pre-specified; ANOVA with fixed factors for study period and treatment, while subject was random effect; Adjusted Mean Difference = 1.60, 95% CI 2-sided [1.36 to 1.85] — [estimate comment as in outcome 3, analysis 3]
Statistical Analysis 5: Comparison: NaF Dentifrice (250 ppmF) vs Placebo Dentifrice (0 ppmF); Null hypothesis considered no difference between treatments, being compared; Test type: Superiority or Other; p < 0.0001, ANOVA — No adjustment was required for multiple comparisons as primary comparison was pre-specified; ANOVA with fixed factors for study period and treatment, while subject was random effect; Adjusted Mean Difference = 0.62, 95% CI 2-sided [0.38 to 0.86] — [estimate comment as in outcome 3, analysis 3]
Statistical Analysis 6: Comparison: NaF Dentifrice (1426 ppmF) vs NaF Dentifrice (1150 ppmF); Null hypothesis considered no difference between treatments, being compared; Test type: Superiority or Other; p = 0.6680, ANOVA — No adjustment was required for multiple comparisons as primary comparison was pre-specified; ANOVA with fixed factors for study period and treatment, while subject was random effect; Adjusted Mean Difference = 0.05, 95% CI 2-sided [-0.19 to 0.29] — [estimate comment as in outcome 3, analysis 3]
Statistical Analysis 7: Comparison: NaF Dentifrice (1426 ppmF) vs NaF Dentifrice (250 ppmF); Null hypothesis considered no difference between treatments, being compared; Test type: Superiority or Other; p < 0.0001, ANOVA — No adjustment was required for multiple comparisons as primary comparison was pre-specified; ANOVA with fixed factors for study period and treatment, while subject was random effect; Adjusted Mean Difference = 1.04, 95% CI 2-sided [0.80 to 1.28] — [estimate comment as in outcome 3, analysis 3]
Statistical Analysis 8: Comparison: NaF Dentifrice (1150 ppmF) vs NaF Dentifrice (250 ppmF); Null hypothesis considered no difference between treatments, being compared; Test type: Superiority or Other; p < 0.0001, ANOVA — No adjustment was required for multiple comparisons as primary comparison was pre-specified; ANOVA with fixed factors for study period and treatment, while subject was random effect; Adjusted Mean Difference = 0.99, 95% CI 2-sided [0.75 to 1.23] — [estimate comment as in outcome 3, analysis 3]

ADVERSE EVENTS:
Time Frame: All adverse events encountered or spontaneously reported following administration of any investigational product (including washout product), or for up to 5 days after the last administration of investigational product were recorded.
Groups:
- NaF Dentifrice (1426 ppmF): Participants brushed their teeth for one timed minute with 1.5 g ± 0.1g of NaF toothpaste (1426 ppmF) and expectorated.
- NaF Dentifrice (1150 ppmF): Participants brushed their teeth for one timed minute with 1.5 g ± 0.1g of NaF toothpaste (1150 ppmF) and expectorated.
- NaF Dentifrice (250 ppmF): Participants brushed their teeth for one timed minute with 1.5 g ± 0.1g of NaF toothpaste (250 ppmF) and expectorated.
- Placebo Dentifrice (0 ppmF): Participants brushed their teeth for one timed minute with 1.5 g ± 0.1g of placebo toothpaste (0 ppmF) and expectorated.
Arm/Group | NaF Dentifrice (1426 ppmF) | NaF Dentifrice (1150 ppmF) | NaF Dentifrice (250 ppmF) | Placebo Dentifrice (0 ppmF)
Serious Adverse Events (participants affected / at risk) | 0/62 | 0/61 | 0/62 | 0/60
Other Adverse Events (participants affected / at risk) | 3/62 | 6/61 | 1/62 | 4/60
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NaF Dentifrice (1426 ppmF) (N=62) | NaF Dentifrice (1150 ppmF) (N=61) | NaF Dentifrice (250 ppmF) (N=62) | Placebo Dentifrice (0 ppmF) (N=60)
Mouth Ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tooth Abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mouth Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tongue Hematoma (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal Pain, Upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sensitivity of teeth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.